CLINICAL TRIAL: NCT01435200
Title: Prevention of Blood Transfusion With Intravenous Iron in Gynecologic Cancer Patients Receiving Platinum Based Chemotherapy
Brief Title: Intravenous Iron in Gynecologic Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Tarinee Manchana, Department of Obstetrics and Gynecology, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IV iron 2
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Gynecologic Cancer
Keywords: Intravenous iron; gynecologic cancer blood transfusion
MeSH Terms: interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous iron (Experimental): Iron sucrose 200 mg intravenous infusion in 15 minutes
  Interventions: Drug: Intravenous iron
- Oral iron (Placebo Comparator): Ferrous fumarate 200 mg oral three times a day
  Interventions: Drug: Intravenous iron

INTERVENTIONS:
Drug: Intravenous iron — Intravenous iron 200 mg add in 0.9% Normal saline 100 ml infused within 15 minutes after every cycles of chemotherapy
  Other Names: Venofer

SUMMARY:
Can intravenous iron lower the rate of blood transfusion in gynecologic cancer patients receiving platinum based chemotherapy than oral iron?

DETAILED DESCRIPTION:
Anemia is a common condition during chemotherapy administration. Treatment options usually include oral iron supplementation and blood transfusion. However, oral iron has gastrointestinal side effects, which affects patient compliance, and only a small amount of oral iron can be absorbed from the gastrointestinal tract. Intravenous iron may overcome a block of iron absorption and iron recycling induced by hepcidin. Therefore, it may increase hemoglobin level and reduced blood transfusion in cancer patients receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-70 years
* Good performance status (Zubrod score < 2)
* No serious underlying disease
* Normal renal function test
* Normal liver function test
* Platinum based chemotherapy is the first line regimen
* No prior or receiving radiotherapy

Exclusion Criteria:

* Iron hypersensitivity
* Underlying disease which has the risk of iron overload such as chronic kidney disease, major thalassemia
* Progressive disease
* Bone marrow metastasis

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Red blood cell (RBC) transfusion rate | 6 months
  The requirement of red blood cell transfusion before administration of chemotherapy will be evaluated for 6 cycles of chemotherapy.

SECONDARY OUTCOMES:
total number of red blood transfusion units and number of cycles requiring blood transfusion | 6 months
Number of participants with adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tarinee Manchana, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Athibovonsuk P, Manchana T, Sirisabya N. Prevention of blood transfusion with intravenous iron in gynecologic cancer patients receiving platinum-based chemotherapy. Gynecol Oncol. 2013 Dec;131(3):679-82. doi: 10.1016/j.ygyno.2013.09.028. Epub 2013 Oct 5. PMID 24099839